CLINICAL TRIAL: NCT00684372
Title: BK Viremia After Renal Transplantation: Screening, Early Diagnosis, Early Reduction in Immunosuppression and Treatment With Leflunomide (Arava)
Brief Title: BK Viremia After Renal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Lars Wennberg, Associate Professor, Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BK study
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Terminal Renal Failure; BK Virus Infection
MeSH Terms: interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: leflunomide — Screening: If BK viremia (BK PCR >10 000 copies/ml in serum) i. Reduced immunosuppression
  1. MMF / AZA withdrawal
  2. CNI reduction
     1. Tacrolimus 5 ng/ml in serum
     2. Cyclosporin 100 ng/ml in serum
  3. Prednisolone to maintenance level
  If effective => continue
  * Stable renal function (P-Krea)
  * >50% reduction in PCR (copies/ml) at 4 weeks after diagnosis
  * Negative PCR at > 3 months after diagnosis
  If failure => add leflunomide
  * Deteriorating renal function (P-Krea) and positive PAD = BK nephropathy
  * <50% reduction in PCR at 4 weeks after diagnosis
  * Positive PCR at >3 months after diagnosis
  Leflunomide dosing:
  ii. Loading dose of 100 mgx1 PO daily for 5 days can be used or the patient can be directly started on iii. Maintenance dose (from day 1 or day 6)
  1. Starting at 20 mgx1 PO daily
  2. Thereafter adjusted between approximately 20-60 mgx1 PO daily according to serum levels of A77 1726 and the clinical situation a. Recommended level of A77 1726 >40 ug/ml

SUMMARY:
Hypothesis: Early detection, and treatment, of BK virus infection after kidney transplantation will prevent BK virus associated kidney transplant injury.

BK virus associated nephropathy (BKVN) is estimated to cause a progressive kidney transplant injury in 1-10% of renal transplant recipients. Diagnostic and monitoring strategies for BKVN is still being developed. Detectable virus in the blood by polymerase change reaction-test (PCR) is predictive of BKVN. Additionally, PCR provides a objective estimate of the degree of infection.

If early detection and treatment of BK virus infection is effective in preventing subsequent kidney transplant injury has not been studied. However, renal injury and dysfunction develops late in the natural course of BKVN and it seems likely that screening in combination with early treatment would be beneficial for long-term transplant survival.

There is no established treatment for BK virus infection. Nevertheless, in kidney transplanted patients diagnosed with BK virus infection, immunosuppression is reduced to allow the patients own immune system to handle the virus. However, reduction of immunosuppression has not been associated with rejection. This indicate that these patients were over-immunosuppressed, predisposing them to BKVN. Therefore, to compare the degree of immunosuppression in BKVN patients (over-immunosuppressed) to other patients (not over-immunosuppressed) could yield interesting information. One possibility would be to quantify these patients specific cellular immune response to BK virus but also to other viruses (T cell reactivity).

Leflunomide (Arava) is an immunosuppressive drug, approved for the treatment of rheumatoid arthritis, and has been used in more than 300,000 patients worldwide. Furthermore, leflunomide has been used safely in humans after clinical kidney and liver transplantation for more than 300 days. In addition to leflunomide's value in preventing rejection, it has been shown to exert inhibitory effects on different viruses. Recently published pilot studies suggest that leflunomide treatment of patients with BKVN significantly reduces the amount of BK virus in blood and prevents recurrence of kidney transplant injury. At Karolinska University Hospital, leflunomide has been used for treatment of BKVN and, in some of the patients, renal function has stabilized and BK virus load has decreased significantly.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing kidney transplantation at Karolinska University Hospital

Exclusion Criteria:

* Absence of informed consent
* Allergy to leflunomide
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Renal function (serum creatinine) | 1 year after diagnosis of BK viremia

SECONDARY OUTCOMES:
Incidence of BK virus associated nephropathy | 1 year after diagnosis of BK viremia

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wennberg, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden